CLINICAL TRIAL: NCT00005519
Title: Prospective Study of Diet and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5039; R03HL061954 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Stroke

SUMMARY:
To examine associations between various dietary elements and the risk of coronary heart disease and stroke.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease is the leading cause of death among residents of the United States. The effect of dietary cholesterol and fat on risk of coronary heart disease (CHD) and stroke has been examined extensively in epidemiologic studies. However, the results from these studies are inconsistent. Furthermore, the association between some other key elements of diet and risk of CHD and stroke has been insufficiently studied in epidemiologic studies.

DESIGN NARRATIVE:

The study examines prospectively the association between: 1) dietary intake of trans-unsaturated fat and the risk of coronary heart disease and 2) dietary intake of total, saturated and unsaturated fats and risk of stroke; 3) dietary intake of vegetable and animal protein and risk of stroke; 4) dietary intake of total and water-soluble fiber and risk of coronary heart disease and stroke; 5) dietary intake of sodium and potassium and risk of coronary heart disease and stroke; 6) dietary intake of vitamin C, carotenoids, vitamin E, and folic acid and the risk of coronary heart disease and stroke; and 7) specific foods, such as fish, beans, fruits, and vegetables and the risk of coronary heart disease and stroke. In addition, the association of baseline serum vitamin A, vitamin C, and folate to the risk of coronary heart disease and stroke will be investigated.

Data from the NHANES1 Epidemiologic Follow-Up Study (NHEFS) will be used to test the hypotheses. The NHEFS is an on-going prospective cohort study being conducted in 14,407 United States men and women aged 25 to 74 years by the National Center for Health Statistics (NCHS). The baseline data, including a 24-hour dietary recall and food frequency questionnaire, as well as important cardiovascular risk factors were collected during 1971-75. The follow-up data were collected during 1982 to 1984, 1986, 1987, and 1992. The follow-up data were obtained by means of an interview, medical records from health care facilities, and death certificates for all decedents. In the study, the investigators will re-code dietary data and calculate dietary nutrients using the ESHA Nutrient Database. They will also analyze the relationship of dietary nutrients and specific foods to risk of CHD and stroke.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He — Tulane University

REFERENCES:
- [Background] He J, Ogden LG, Bazzano LA, Vupputuri S, Loria C, Whelton PK. Risk factors for congestive heart failure in US men and women: NHANES I epidemiologic follow-up study. Arch Intern Med. 2001 Apr 9;161(7):996-1002. doi: 10.1001/archinte.161.7.996. PMID 11295963
- [Background] Bazzano LA, He J, Ogden LG, Loria C, Vupputuri S, Myers L, Whelton PK. Legume consumption and risk of coronary heart disease in US men and women: NHANES I Epidemiologic Follow-up Study. Arch Intern Med. 2001 Nov 26;161(21):2573-8. doi: 10.1001/archinte.161.21.2573. PMID 11718588
- [Background] He J, Ogden LG, Vupputuri S, Bazzano LA, Loria C, Whelton PK. Dietary sodium intake and subsequent risk of cardiovascular disease in overweight adults. JAMA. 1999 Dec 1;282(21):2027-34. doi: 10.1001/jama.282.21.2027. PMID 10591385
- [Background] Bazzano LA, He J, Ogden LG, Loria C, Vupputuri S, Myers L, Whelton PK. Dietary potassium intake and risk of stroke in US men and women: National Health and Nutrition Examination Survey I epidemiologic follow-up study. Stroke. 2001 Jul;32(7):1473-80. doi: 10.1161/01.str.32.7.1473. PMID 11441188